CLINICAL TRIAL: NCT01794208
Title: A Phase II, Multicentre, Multinational, Randomised, Assessor-Blind Trial to Investigate the Efficacy and Safety of Various Dosages of FSH-GEX™ in Comparison With 150 IU Gonal-f® in Women Undergoing ICSI Treatment
Brief Title: Efficacy and Safety of FSH-GEX™ in Comparison With 150 IU Gonal-f®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glycotope GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GEXGP24201
Record Dates: First submitted 2013-01-23; First posted 2013-02-18 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Infertility
Keywords: in-vitro fertilization; reproductive disorder
MeSH Terms: conditions — Infertility | interventions — follitropin alfa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (6):
- treatment 1 (Experimental): Follitropin Epsilon 52.5 IU quaque die (QD) s.c.
  Interventions: Drug: Follitropin Epsilon
- treatment 2 (Experimental): Follitropin Epsilon 75 IU QD s.c.
  Interventions: Drug: Follitropin Epsilon
- treatment 3 (Experimental): Follitropin Epsilon 112.5 IU QD s.c.
  Interventions: Drug: Follitropin Epsilon
- treatment 4 (Experimental): Follitropin Epsilon 150 IU QD s.c.
  Interventions: Drug: Follitropin Epsilon
- treatment 5 (Experimental): Follitropin Epsilon 150 IU quaque altera die (QAD) s.c.
  Interventions: Drug: Follitropin Epsilon
- treatment 6 (Active Comparator): Follitropin alfa 150 IU QD s.c.
  Interventions: Drug: Follitropin Alfa

INTERVENTIONS:
Drug: Follitropin Epsilon
  Other Names: FSH-GEX(TM)
  Arms: treatment 1; treatment 2; treatment 3; treatment 4; treatment 5
Drug: Follitropin Alfa
  Other Names: Gonal-f(R)
  Arms: treatment 6

SUMMARY:
The aim of the current study was the determination of the recommended standard treatment dose of FSH-GEX(TM) in women undergoing intracytoplasmic sperm injection (ICSI) treatment as assessed by follicle growth.

DETAILED DESCRIPTION:
This was a phase II, randomized, assessor-blind, comparator-controlled, multiple dose study in women undergoing ICSI treatment.

The primary objective of the study was the determination of the recommended standard treatment dose of FSH-GEX™ as assessed by follicle growth dynamics in women between 18 and 37 years of age who were undergoing intracytoplasmic sperm injection treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patient for whom ICSI treatment is justified
* Serum follicle-stimulating hormone concentration
* Anti-mullerian hormone concentration
* Antral follicle count
* Body mass index and body weight
* Presence of both ovaries
* Regular spontaneous cycles between 21 and 35 days in length
* Normal uterine cavity as assessed by transvaginal sonography at Screening
* Willing and able to comply with the protocol
* Willing and able to provide written informed consent

Exclusion Criteria:

* Patients who had more than two unsuccessful previous assisted reproduction technology cycles before inclusion into the study
* Previous poor responders
* Patients with previous hyperstimulation syndrome or cycle cancellation because of imminent hyperstimulation syndrome
* Patients with a history of or current polycystic ovarian morphology syndrome
* Patients with a history of or current endometriosis III or IV
* Presence of ovarian cyst at Screening
* Any contraindication to becoming pregnant
* History of ≥ 3 clinical or preclinical miscarriages
* Abnormal cervical smear, Papanicolaou [PAP] score ≥ 3
* Any history of malignant cancer other than in situ breast or skin cancer requiring local excision
* Any endocrine abnormalities requiring treatment
* Any clinically significant systematic disease
* Any known infection with human immunodeficiency virus, hepatitis B or C
* History of thrombosis or other risk factors including any coagulation abnormality leading to an increased risk of clotting
* Family history of genetic risk factors concerning pregnancy or birth
* Use of concomitant medication, which in the opinion of the investigator might interfere with ICSI preparation procedures
* Active smoking
* Any active substance abuse of drugs, medications or alcohol within the last five years
* Patients in an institution by official or court order
* Patients who are unable or unwilling to provide informed consent
* Any participation in another clinical trial within the last 60 days before randomisation
* Previous FSH-GEX™ administration.
* Known hypersensitivity to any component of the investigational and non investigational products used in this study

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 267 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07-30 (Actual)

PRIMARY OUTCOMES:
Number of follicles | day of hCG injection; variable timeframe; up to 18 days for maximum
  The number of follicles with a diameter of ≥ 12 mm on the day of human chorionic gonadotropin (hCG) injection after stimulation with follicle stimulating hormone (FSH)

SECONDARY OUTCOMES:
Follicular response | every second day up to hCG injection; variable timeframe; up to 18 days for maximum
  For each ovary the number of follicles were classified and summarised as follows: mean diameter 8.0 - 9.9 mm, 10.0 - 11.9 mm, 12.0 - 13.9 mm, 14.0 - 15.9 mm, 16.0 - 17.9 mm, 18.0 - 19.9 mm, and >19.9 mm as determined by transvaginal ultrasonography
Cumulus-oocyte-complexes | at oocyte retrieval; 32 - 36 hours after hCG injection
  Number of retrieved cumulus-oocyte-complexes
Oocytes retrieved | at oocyte retrieval; 32 - 36 hours after hCG injection
  Number of oocytes retrieved (metaphase II)
Two pronuclei oocytes | one day after oocyte retrieval
  Number of two pronuclei (2PN) oocytes one day after follicle puncture
Biochemical pregnancy rate | 14 to 20 days after oocyte retrieval
  Based on positive β-hCG pregnancy test
Clinical pregnancy rate | approx. 4 to 6 weeks after last FSH dose
  Based on clinical or ultrasound parameters (gestational sac, foetal heart beat
Implantation rate | approx. 4 to 6 weeks after last FSH dose
  Number of foetal sacs on sonography divided by number of embryos transferred per embryo transfer
Estradiol and inhibin B serum levels | every second day up to hCG injection; variable timeframe; up to 18 days maximum
  Concentration of Estradiol and Inhibin B in Serum after FSH stimulation
Adverse events, ovarian hyperstimulation syndrome, anti-drug-antibodies, overall tolerability | up to 4 to 6 weeks after last FSH dose
  Incidence of adverse events, ovarian hyperstimulation syndrome, anti-drug-antibodies, overall tolerability
Number of doses and total dose of FSH | variable timeframe; up to 18 days for maximum
  The total dose is the amount of FSH-GEX(TM) or Gonal-f® administered to each patient during the stimulation period

OTHER OUTCOMES:
Ongoing pregnancy rate | 10 weeks after gestation
  A pregnancy is considered an ongoing pregnancy if pregnancy can be confirmed for more than 10 weeks after gestation.
Life birth rate | up to nine month after embryo transfer
  The live birth rate will be calculated as the total number of live births divided by the number of randomised patients

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Glycotope GmbH
Locations (7):
- Germany (5):
  - Glycotope Investigational Site, Berlin
  - Glycotope Investigational Medical Director, Bielefeld
  - Glycotope Investigational Site, Düsseldorf
  - Glycotope Investigational Site, Heidelberg
  - Glycotope Investigational Site, Lübeck
- Hungary (2):
  - Glycotope Investigational Site, Budapest
  - Glycotope Investigational Site, Tapolca

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Griesinger G, Dietrich B, Stockl L, Eckert K, Goletz S, Tandler-Schneider A. Fully human glyco-optimized recombinant FSH (follitropin epsilon) - a randomized, comparator-controlled phase II clinical trial. Reprod Biomed Online. 2020 Feb;40(2):331-341. doi: 10.1016/j.rbmo.2019.09.003. Epub 2019 Sep 16. PMID 31982355